CLINICAL TRIAL: NCT07065435
Title: Efficacy and Safety of Disitamab Vedotin (RC48) in Combination With Bevacizumab or Pyrotinib in Patients With HER2-Positive Metastatic Breast Cancer After Trastuzumab Deruxtecan (T-DXd) Treatment Failure: A Phase II Study
Brief Title: RC48 Plus Bevacizumab or Pyrotinib in HER2-Positive Metastatic Breast Cancer After T-DXd Failure: A Phase II Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: RenJi Hospital (Other); Anhui Provincial Hospital (Other Government); The Affiliated Hospital of Xuzhou Medical University (Other); The First Hospital of Jilin University (Other); Shanghai Minhang Central Hospital (Other); Zhejiang Cancer Hospital (Other); Huai'an First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJMU-BC07
Record Dates: First submitted 2025-07-02; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: HER2 + Breast Cancer
Keywords: Disitamab Vedotin (RC48); Bevacizumab; Pyrotinib; Trastuzumab deruxtecan failure
MeSH Terms: conditions — Breast Neoplasms | interventions — disitamab vedotin; RC48 antibody; Bevacizumab; pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RC48 + Bevacizumab (Experimental): Participants receive Disitamab Vedotin (RC48) at 2.0 mg/kg IV every 2 weeks plus Bevacizumab 7.5 mg/kg IV every 2 weeks. Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or initiation of new anticancer therapy.
  Interventions: Drug: Disitamab Vedotin (RC48); Drug: Bevacizumab
- RC48 + Pyrotinib (Experimental): Participants receive Disitamab Vedotin (RC48) at 2.0 mg/kg IV every 2 weeks plus Pyrotinib 320 mg orally once daily (post-meal). Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or initiation of new anticancer therapy.
  Interventions: Drug: Disitamab Vedotin (RC48); Drug: Pyrotinib

INTERVENTIONS:
Drug: Disitamab Vedotin (RC48) — A HER2-targeted antibody-drug conjugate comprising a humanized anti-HER2 monoclonal antibody linked via a cathepsin-cleavable MC-VC-PAB linker to the microtubule inhibitor MMAE (drug-to-antibody ratio ≈4). Administered intravenously at 2.0 mg/kg every 2 weeks.
Drug: Bevacizumab — A recombinant humanized monoclonal antibody that binds vascular endothelial growth factor (VEGF) to inhibit tumor angiogenesis. Administered intravenously at 7.5 mg/kg every 2 weeks in combination with RC48.
  Arms: RC48 + Bevacizumab
Drug: Pyrotinib — An irreversible pan-HER tyrosine kinase inhibitor targeting HER1, HER2, and HER4, inhibiting downstream PI3K/Akt and MAPK signaling. Administered orally at 320 mg once daily (post-meal) in combination with RC48.
  Arms: RC48 + Pyrotinib

SUMMARY:
This multicenter, Phase II study (RADIANT-BC01) evaluates the efficacy and safety of Disitamab Vedotin (RC48) in combination with either bevacizumab or pyrotinib in adult patients with HER2-positive metastatic breast cancer whose disease has progressed on prior trastuzumab deruxtecan (T-Dxd) therapy.

Eligible participants will be randomized 1:1 to receive RC48 plus bevacizumab (7.5 mg/kg IV every 2 weeks) or RC48 plus pyrotinib (320 mg orally once daily). Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or initiation of new anticancer therapy.

The primary endpoint is objective response rate (ORR); key secondary endpoints include progression-free survival (PFS), disease control rate (DCR), duration of response (DOR), overall survival (OS), and safety.

This study aims to identify new post-T-Dxd treatment options and improve outcomes for patients with advanced HER2-positive breast cancer.

DETAILED DESCRIPTION:
Despite the remarkable benefits of trastuzumab deruxtecan (T-Dxd) as second-line therapy, resistance inevitably develops in HER2-positive metastatic breast cancer, and no standard treatment exists after T-Dxd failure. Disitamab Vedotin (RC48) is a novel antibody-drug conjugate (ADC) targeting HER2, with a cathepsin-cleavable linker and MMAE payload that has demonstrated encouraging antitumor activity and tolerability in earlier studies. Preclinical and real-world data suggest that combining RC48 with anti-angiogenic agents (bevacizumab) or a pan-HER tyrosine kinase inhibitor (pyrotinib) may enhance tumor penetration, overcome resistance mechanisms, and provide synergistic effects without overlapping toxicity.

RADIANT-BC01 is designed as two parallel Simon two-stage cohorts: one evaluating RC48 + bevacizumab and the other RC48 + pyrotinib. In each arm, 14 patients will be enrolled in the first stage, with progression to a total of 37 patients if at least five responses are observed. Patients must have received at least two cycles of prior T-Dxd, possess measurable disease per RECIST 1.1, an ECOG performance status of 0-2, and adequate organ function. Key exclusion criteria include uncontrolled comorbidities, active interstitial lung disease, and prior adverse reactions to study agents.

The study's primary objective is to determine the ORR of each combination regimen. Secondary objectives encompass PFS, DCR, DOR, OS, and safety assessments. Exploratory biomarker analyses will be conducted on serial blood and stool samples to identify predictors of response and resistance. Tumor assessments occur every 6 weeks, with safety evaluations at each treatment visit and a follow-up period of 90 days post-treatment, then every 3 months for survival status. By exploring these combination strategies, RADIANT-BC01 seeks to establish new therapeutic options for patients who have exhausted current HER2-targeted treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically or cytologically confirmed HER2-positive (IHC 3+ or IHC 2+ with ISH amplification) advanced or metastatic breast cancer.
3. Prior treatment with trastuzumab deruxtecan (T-DXd) and documented disease progression during or after therapy.
4. At least one measurable lesion at baseline as defined by RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Adequate organ and marrow function, including:

Absolute neutrophil count ≥1.5 × 10⁹/L Platelet count ≥100 × 10⁹/L Hemoglobin ≥9 g/dL ALT and AST ≤2.5 × ULN Total bilirubin ≤1.5 × ULN Creatinine clearance ≥50 mL/min Estimated life expectancy of ≥12 weeks. Ability to understand and willingness to sign a written informed consent form.

Exclusion Criteria:

1. Prior treatment with disitamab vedotin (RC48).
2. Active infections requiring systemic therapy (bacterial, viral, or fungal).
3. History of interstitial lung disease or non-infectious pneumonitis requiring corticosteroid therapy.
4. Uncontrolled cardiovascular disease, including but not limited to: uncontrolled hypertension, recent myocardial infarction (within 6 months), unstable angina, or congestive heart failure.
5. Pregnant or breastfeeding women.
6. Concurrent malignancy other than adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix, unless disease-free for ≥5 years.
7. Participation in another interventional clinical trial with investigational agents not yet completed.
8. Any condition that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements or jeopardize their safety.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The Objective Response Rate (ORR) is defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) according to RECIST version 1.1 criteria, as assessed by independent radiological review. Tumor assessments will be performed every 6 weeks. This endpoint evaluates the antitumor activity of RC48 in combination with either bevacizumab or pyrotinib in patients with HER2-positive advanced breast cancer who have failed prior treatment with trastuzumab deruxtecan (T-Dxd).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-Free Survival is defined as the time from the date of randomization to the date of first documented disease progression (per RECIST v1.1 by independent review) or death from any cause, whichever occurs first. PFS will be used to evaluate the efficacy of the combination regimens in delaying disease progression in patients with HER2-positive advanced breast cancer previously treated with trastuzumab deruxtecan.
Overall Survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall Survival is defined as the time from randomization to death from any cause. Patients who are still alive at the time of analysis will be censored at the date of last follow-up. OS will provide a measure of the survival benefit of RC48 combined with either bevacizumab or pyrotinib.
Duration of Response (DoR) | From first documented response until disease progression or death, assessed up to 24 months
  Duration of Response is defined as the time from the first documentation of objective tumor response (CR or PR per RECIST v1.1) to the time of disease progression or death. Only patients with confirmed objective response will be included in this analysis.
Disease Control Rate (DCR) | Assessed at 6 weeks and every 8 weeks thereafter up to 24 months
  Disease Control Rate is defined as the proportion of patients who achieve a complete response (CR), partial response (PR), or stable disease (SD) lasting at least 6 weeks, based on RECIST v1.1 as assessed by independent review.
Incidence of Treatment-Related Adverse Events | From first dose until 30 days after last dose, assessed up to 36 months
  The incidence and severity of treatment-related adverse events (TRAEs) will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. This measure aims to evaluate the safety and tolerability of the treatment regimens.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code